CLINICAL TRIAL: NCT01780597
Title: Ex Vivo Assessment of Human Hearts Deemed Unsuitable for Cardiac Transplant With the Ultimate Aim of Increasing the Number of Hearts Available for Transplant for Cardiac Failure Patients.
Brief Title: Assessment of Hearts Deemed Unsuitable for Transplant With the Aim of Expanding the Donor Heart Pool.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: NewcastleNHS
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure
Keywords: Heart transplantation; Ev Vivo Perfusion; Cardiac function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocardial biopsies, serum samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Organ Donors (declared Brainstem-Dead): This group of subjects is defined as those who have previously expressed their future wish to organ donation and who have suffered events leading to declaration of brainstem-death. Furthermore these subjects will have had their hearts declined for heart transplantation on the basis of poor function.

SUMMARY:
The main question to be asked in this study is what is the potential for human hearts that have been deemed unacceptable for transplant, to be explanted and re-animated in a controlled, external environment to be assessed? Furthermore would the reanimated hearts be able to undergo improvement in their function in this external environment.

Ultimately this may lead to an increase the number of hearts available for transplantation.

DETAILED DESCRIPTION:
Year on year with improvement in road safety and improvement in neurosurgery the number of ideal young brain dead donors have been declining whilst the number of more marginal donors have been increasing. The consequence of this is the number of heart transplants being performed have steadily declined.

At present there are 600 hearts from brain dead donors offered for transplant every year in the United Kingdom (UK). Of these 200 have anatomical reasons why they cannot be used for transplant such as ischaemic heart disease. 100 are transplanted and the remaining 300 hearts are judged to have inferior function which probably occurs as a direct result of brain death (Dark).

Ex vivo 'rig' testing has been developed for lungs that were judged unsuitable for transplantation. As a result several donor lungs have been 'improved' by warm perfusion on the rig to the extent that they became suitable for transplantation and so national lung transplant rates are increasing (Dark). The aim would be to develop a similar approach for the heart.

ELIGIBILITY:
Inclusion Criteria:

* Participant is brain dead and their relative is willing to give informed consent
* Male or Female, aged between 18 and 75 years
* Heart is not eligible for transplantation

Exclusion Criteria:

* Participant's relative refuses consent
* Brain dead donor whose heart is eligible for transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organ Donors (declared brainstem dead). The hearts are only to be studied after death and removal from the body. Consent given first from the next of kin.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2013-02; Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
The investigators aim to measure an improvement in cardiac function (ie contractility) by measuring the Pressure Change/Time max (dP/dT), in mmHg/second, of the heart once it has achieved reanimation on the ex vivo circuit. | 12 hours
  Can human hearts that have been deemed unacceptable for transplant be re-animated in a controlled, external environment to be assessed? Furthermore, can their function (contractility) be improved by ex vivo reperfusion? This will be measured using conductance catheters to measure the dP/dT max (mmHg/second) at various time intervals.

SECONDARY OUTCOMES:
Can their function (contractility measured in mmHg/second) of the hearts be improved by an additional re-oxygenation step during the cold phase of heart preservation? | 24 hours
  Can these hearts be improved during the cold phase of transportation by either continuous circulation of preservation solution or oxygen gas through the heart? Hearts will be reperfused on the ex vivo circuit having been subjected to either method of preservation and their contractility measurements (mmHg/sec) once reanimated will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: David Talbot, MBBS PhD MD, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Freeman Hospital, Newcastle upon Tyne, Tyne & Wear, United Kingdom

REFERENCES:
- [Background] Botha P, MacGowan GA, Dark JH. Sildenafil citrate augments myocardial protection in heart transplantation. Transplantation. 2010 Jan 27;89(2):169-77. doi: 10.1097/TP.0b013e3181c42b22. PMID 20098279
- [Background] Dark JH. Lung transplantation from the non-heart beating donor. Transplantation. 2008 Jul 27;86(2):200-1. doi: 10.1097/TP.0b013e31817c87b6. PMID 18645477
- [Background] Macgowan GA, Parry G, Schueler S, Hasan A. The decline in heart transplantation in the UK. BMJ. 2011 May 5;342:d2483. doi: 10.1136/bmj.d2483. No abstract available. PMID 21546420
- [Background] Redfield MM. Heart failure--an epidemic of uncertain proportions. N Engl J Med. 2002 Oct 31;347(18):1442-4. doi: 10.1056/NEJMe020115. No abstract available. PMID 12409548